CLINICAL TRIAL: NCT02230085
Title: A Validation Study of an Adherence Risk Indicator Statistical Prediction Model.
Brief Title: Adherence Risk Indicator Validation Study
Acronym: ARI
Status: Completed | Type: Observational
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: CIA-121
Record Dates: First submitted 2014-08-19; First posted 2014-09-03 (Estimated); Results first posted 2016-12-02 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CPAP therapy
  Interventions: Other: Administration of the questionnaire and monitoring of CPAP adherence

INTERVENTIONS:
Other: Administration of the questionnaire and monitoring of CPAP adherence

SUMMARY:
While continuous positive airway pressure (CPAP) is the gold standard treatment of obstructive sleep apnea (OSA), this therapy is often discontinued or not used optimally. The adherence risk indicator (ARI) is a statistical model based on answers from a questionnaire. The data collected from this trail allows for closer monitoring of at-risk patients. For the study, participants are provided with a questionnaire prior to starting CPAP therapy for OSA. Participants will be provided with a GSM (Global System for Mobile communication) modem to allow transmission of their CPAP data. Participants data will be retrieved at 7, 14, 21, 30 and 90 days to test the accuracy of the ARI prediction. At the conclusion of the study the GSM unit is returned, and participants continue with CPAP therapy as instructed by their healthcare provider.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18years of age
* Diagnosed with OSA (AHI >5 events/hour) and eligible for CPAP (fixed or auto) treatment under local requirements
* Naïve to CPAP therapy, i.e. have not been prescribed CPAP in the past 5 years

Exclusion Criteria:

* Contraindicated for CPAP therapy
* Medically unstable condition/diagnosis that is not yet under control
* Co-existing sleep disorder (however clinically diagnosed insomnia can be included in the study)
* PLMA (Periodic Limb Movement Activity) Index greater than 15/hr
* Home titration of longer than 5 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient recieving CPAP for OSA.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- EverythingCPAP, Boise, Idaho, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CPAP Therapy: Administration of the questionnaire and monitoring of CPAP adherence
Period: Overall Study
Arm/Group | CPAP Therapy
Started | 110
Completed | 106
Not Completed | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | CPAP Therapy
Number analyzed (Participants) | 103
Age, Continuous [Mean (Full Range); unit: years] | 51 [27 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 60
Region of Enrollment [Number; unit: participants]
  United States | 103

OUTCOME MEASURES:

1. Primary Outcome: CPAP Therapy Adherence
Description: Adherence is measured by the amount of CPAP use (e.g. good adherence was defined as use of greater than or equal to 70% of nights for greater than 4 hours per night). CPAP data was remotely collected and analyzed from the data reports generated by data collection.
Time Frame: 90 days
Population: 103 patients CPAP therapy adherence data was collected. 3 patients data was either lost or unable to be downloaded.
Measure: Number; unit: participants
Arm/Group | CPAP Therapy
Number analyzed (Participants) | 103
participants | 103

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 90 days for each participant.
Arm/Group | CPAP Therapy
All-Cause Mortality (participants affected / at risk) | 0/110
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 0/110

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for an undescribed period .